CLINICAL TRIAL: NCT01215292
Title: Mechanisms of Control of the Intratesticular Hormonal Milieu in Man
Brief Title: ITT4 Intratesticular Hormonal Milieu in Man (ITT4)
Acronym: ITT4
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Mara Roth, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38692-K; U54HD012629 (NIH)
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2014-01-29 (Estimated); Last update posted 2014-03-31 (Estimated); Status verified 2014-02

CONDITIONS: Healthy Males
Keywords: testosterone; acyline; ketoconazole; dutasteride; anastrazole; Intratesticular hormone concentration
MeSH Terms: interventions — acyline; Testosterone; Dutasteride; Anastrozole

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- Acyline & T Gel & Placebo Ketoconazole (Placebo Comparator): Acyline 300 mcg/kg on Day 1 + 1% testosterone gel (T gel) 5 gm daily Days 1-10, + placebo tab PO 1x daily, Day 3-10
  Interventions: Drug: Acyline; Drug: Testosterone gel; Drug: Placebo ketoconazole
- Acyline & T Gel & Ketoconazole 400 (Experimental): Acyline 300 mcg/kg on Day 1 + 1% testosterone gel 5 gm daily Days 1-10, + ketoconazole 400mg PO 1x daily, Days 3-10
  Interventions: Drug: Acyline; Drug: Testosterone gel; Drug: ketoconazole 400
- Acyline & T gel & Ketoconazole 800 (Experimental): Acyline 300 mcg/kg on Day 1 + 1% testosterone gel 5 gm daily Day 1-10, + ketoconazole 800mg PO 1x daily, Days 3-10
  Interventions: Drug: Acyline; Drug: Testosterone gel; Drug: Ketoconazole 800
- Acyline & T gel & Dutasteride (Experimental): Acyline 300 mcg/kg on Day 1 + 1% testosterone gel 5 gm daily Day 1-10, + dutasteride 2.5 mg PO 1x daily, Days 3-10
  Interventions: Drug: Acyline; Drug: Testosterone gel; Drug: Dutasteride
- Group 5: anastrazole (Experimental): Acyline 300 mcg/kg on Day 1 + 1% testosterone gel 5 gm daily Day 1-10, + anastrazole 1 mg PO 1x daily, Days 3-10
  Interventions: Drug: Acyline; Drug: Testosterone gel; Drug: Anastrozole

INTERVENTIONS:
Drug: Acyline — 300 mcg/kg on Day 1
  Other Names: Acyline GnRH antagonist
Drug: Testosterone gel — 5 gm of 1% T Gel applied transdermally for 10 days
  Other Names: Androgel
Drug: ketoconazole 400 — 400 mg PO daily, Days 3-10
  Other Names: Teva
  Arms: Acyline & T Gel & Ketoconazole 400
Drug: Ketoconazole 800 — 800 mg PO daily, Day 3-10
  Other Names: Teva
  Arms: Acyline & T gel & Ketoconazole 800
Drug: Dutasteride — 2.5 mg PO daily, Day 3-10
  Other Names: Avodart
  Arms: Acyline & T gel & Dutasteride
Drug: Anastrozole — 1 mg PO daily, Day 3-10
  Other Names: Arimidex
  Arms: Group 5: anastrazole
Drug: Placebo ketoconazole — placebo to mimic ketoconazole
  Arms: Acyline & T Gel & Placebo Ketoconazole

SUMMARY:
The purpose of this research study is to determine how much male hormone, testosterone, is necessary to maintain sperm production in the testis. This knowledge will be used to help in the development of a safe male hormonal contraception.

Specific Aims:

1. to determine if ketoconazole plus acyline will suppress intratesticular testosterone(ITT) to a greater degree than acyline alone.
2. to determine if dutasteride plus acyline will suppress intratesticular dihydrotestosterone (IT-DHT) to a greater degree than acyline alone.
3. to determine if anastrazole plus acyline will suppress intratesticular estradiol(IT-E2) to a greater degree than acyline alone.

DETAILED DESCRIPTION:
Five drugs will be used in this study: acyline, testosterone gel, ketoconazole, dutasteride, and anastrazole.

Acyline suppresses luteinizing hormone (LH) and follicle stimulating hormone (FSH), which are hormones made by the pituitary gland in the brain, thus blocking the signal from the brain that causes the testes to make testosterone. Therefore, acyline blocks testosterone production. Men may experience some side effects from the low levels of testosterone caused by acyline. Acyline is an experimental drug. Over 125 men have received acyline from our lab. Acyline will be given by injection, and injections are formulated by subject's weight and may be given in multiple injections.

Testosterone gel is given to replace testosterone level back to the normal range. Testosterone gel is approved for use in men with low testosterone levels.

Ketoconazole suppresses testosterone production as well. Ketoconazole works in the adrenal glands to prevent testosterone production. It is approved by the U.S. FDA for treatment of fungal infections but for this study the use is considered investigational.

Dutasteride blocks metabolism of testosterone into dihydrotestosterone (DHT). It is approved by the FDA for treatment of benign enlargement of the prostate gland, but the use is considered investigational in this study. Also, the dose is 5 times higher than the FDA approved dose.

Anastrazole blocks metabolism of testosterone into estradiol. It is approved by the FDA for treatment of breast cancer but its use is considered investigational in this study.

Participation will last approximately 2 months. The study involves a minimum of 7 visits. Clinic visits at Screening, Day 3 and Day 10 will take about 1-1.5 hours each. On Day 3 & 10 a fine needle aspiration of one testis will be performed. The Day 1 visit will take approximately 45 minutes. The Day 7 visit will take about 15 minutes. The Day 17 and Day 40 visits will take approximately 30 minutes each. Over the course of the study, which includes 7 separate blood draws, approximately 12 ounces (one and a half cups) of blood will be drawn. The acyline will be given by injection. The testosterone or placebo gel is applied to the skin on the chest, upper arms, and upper back. The ketoconazole, dutasteride, anastrazole, or placebo medication will be taken by mouth.

Subjects randomly assigned to Group 3 will have a Cosyntropin Stimulation Test performed at the day 10 visit to evaluate the function of adrenal glands.

This is NOT a trial of a male contraceptive, and the study medications will not prevent pregnancy. Subjects must use an acceptable form of birth control.

ELIGIBILITY:
INCLUSION CRITERIA:

* Males age 18-50
* Normal serum testosterone, LH and FSH
* prostate-specific antigen (PSA) < 4.0
* Agrees not to donate blood or participate in another research study during the study
* Informed consent
* Able to understand and comply with protocol requirements, instructions and protocol-stated restrictions
* In general good health based on normal screening evaluation (consisting of a medical history, physical exam, normal serum chemistry and hematology)
* Must be willing to use a reliable form of contraception during the study

EXCLUSION CRITERIA:

* Poor general health, with clinically significant abnormal blood results
* Participation in a long-term male contraceptive study within the past three months
* Participation in long-term contraceptive or drug study within the past 3 months
* History of or current liver disease
* Current use of terfenadine, astemizole, cisapride, budesonide, felodipine, fluticasone, lovastatin, midazolam, sildenafil, or vardenafil
* History of testicular, prostate, or scrotal surgery/trauma or genital abnormal exam
* BMI > 32
* History of sleep apnea and/or major psychiatric problems
* Chronic pain syndrome
* History of testosterone or anabolic steroid abuse currently or in the past
* Known bleeding disorder or current use of anticoagulation
* History of or current skin disorder that will interfere with testosterone gel
* Unwilling to adhere to protocol-stated restrictions while in the study

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mara Y Roth, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Background] Contraceptive efficacy of testosterone-induced azoospermia in normal men. World Health Organization Task Force on methods for the regulation of male fertility. Lancet. 1990 Oct 20;336(8721):955-9. PMID 1977002
- [Background] Wu FC, Farley TM, Peregoudov A, Waites GM. Effects of testosterone enanthate in normal men: experience from a multicenter contraceptive efficacy study. World Health Organization Task Force on Methods for the Regulation of Male Fertility. Fertil Steril. 1996 Mar;65(3):626-36. PMID 8774299
- [Background] Anawalt BD, Bebb RA, Bremner WJ, Matsumoto AM. A lower dosage levonorgestrel and testosterone combination effectively suppresses spermatogenesis and circulating gonadotropin levels with fewer metabolic effects than higher dosage combinations. J Androl. 1999 May-Jun;20(3):407-14. PMID 10386821
- [Background] Zirkin BR, Santulli R, Awoniyi CA, Ewing LL. Maintenance of advanced spermatogenic cells in the adult rat testis: quantitative relationship to testosterone concentration within the testis. Endocrinology. 1989 Jun;124(6):3043-9. doi: 10.1210/endo-124-6-3043. PMID 2498065
- [Background] Coviello AD, Matsumoto AM, Bremner WJ, Herbst KL, Amory JK, Anawalt BD, Sutton PR, Wright WW, Brown TR, Yan X, Zirkin BR, Jarow JP. Low-dose human chorionic gonadotropin maintains intratesticular testosterone in normal men with testosterone-induced gonadotropin suppression. J Clin Endocrinol Metab. 2005 May;90(5):2595-602. doi: 10.1210/jc.2004-0802. Epub 2005 Feb 15. PMID 15713727
- [Background] Roth MY, Lin K, Amory JK, Matsumoto AM, Anawalt BD, Snyder CN, Kalhorn TF, Bremner WJ, Page ST. Serum LH correlates highly with intratesticular steroid levels in normal men. J Androl. 2010 Mar-Apr;31(2):138-45. doi: 10.2164/jandrol.109.008391. Epub 2009 Sep 24. PMID 19779211
- [Background] Trachtenberg J, Zadra J. Steroid synthesis inhibition by ketoconazole: sites of action. Clin Invest Med. 1988 Feb;11(1):1-5. PMID 2966691
- [Background] Nashan D, Knuth UA, Weidinger G, Nieschlag E. The antimycotic drug terbinafine in contrast to ketoconazole lacks acute effects on the pituitary-testicular function of healthy men: a placebo-controlled double-blind trial. Acta Endocrinol (Copenh). 1989 May;120(5):677-81. doi: 10.1530/acta.0.1200677. PMID 2499150
- [Background] Pont A, Graybill JR, Craven PC, Galgiani JN, Dismukes WE, Reitz RE, Stevens DA. High-dose ketoconazole therapy and adrenal and testicular function in humans. Arch Intern Med. 1984 Nov;144(11):2150-3. PMID 6093722
- [Background] Van Tyle JH. Ketoconazole. Mechanism of action, spectrum of activity, pharmacokinetics, drug interactions, adverse reactions and therapeutic use. Pharmacotherapy. 1984 Nov-Dec;4(6):343-73. doi: 10.1002/j.1875-9114.1984.tb03398.x. PMID 6151171
- [Background] Soriano-Guillen L, Lahlou N, Chauvet G, Roger M, Chaussain JL, Carel JC. Adult height after ketoconazole treatment in patients with familial male-limited precocious puberty. J Clin Endocrinol Metab. 2005 Jan;90(1):147-51. doi: 10.1210/jc.2004-1438. Epub 2004 Nov 2. PMID 15522928
- [Background] Harris KA, Weinberg V, Bok RA, Kakefuda M, Small EJ. Low dose ketoconazole with replacement doses of hydrocortisone in patients with progressive androgen independent prostate cancer. J Urol. 2002 Aug;168(2):542-5. PMID 12131305
- [Background] Herbst KL, Coviello AD, Page S, Amory JK, Anawalt BD, Bremner WJ. A single dose of the potent gonadotropin-releasing hormone antagonist acyline suppresses gonadotropins and testosterone for 2 weeks in healthy young men. J Clin Endocrinol Metab. 2004 Dec;89(12):5959-65. doi: 10.1210/jc.2003-032123. PMID 15579744
- [Result] Roth MY, Nya-Ngatchou JJ, Lin K, Page ST, Anawalt BD, Matsumoto AM, Marck BT, Bremner WJ, Amory JK. Androgen synthesis in the gonadotropin-suppressed human testes can be markedly suppressed by ketoconazole. J Clin Endocrinol Metab. 2013 Mar;98(3):1198-206. doi: 10.1210/jc.2012-3527. Epub 2013 Jan 24. PMID 23348398

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy men, aged 18-50 years were recruited for this study using newspaper and online advertisement, including flyers posted at the University of Washington, Seattle.
Pre-assignment Details: Fifty-two men were screened for the study and 46 met all inclusion criteria. Six subjects withdrew from the study prior to any procedures and 40 were randomized (n=8/group. Exclusion criteria included liver disease or adrenal insufficiency, Body Mass Index > 32, abnormal test results, skin conditions for gel, alcohol/drug abuse etc.
Period: Overall Study
Arm/Group | Acyline & T Gel & Ketoconazole 400 | Acyline & T Gel & Dutasteride | Acyline & T Gel & Placebo Ketoconazole | Acyline & T Gel & Ketoconazole 800 | Group 5: Anastrazole
Started | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Fifty two men were screened for the study and 46 met all inclusion criteria. Six subject withdrew from the study prior to any procedures and 40 were randomized to treatment 8/group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acyline & T Gel & Ketoconazole 400 | Acyline & T Gel & Dutasteride | Acyline & T Gel & Placebo Ketoconazole | Acyline & T Gel & Ketoconazole 800 | Group 5: Anastrazole | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8 | 40
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 22.5 [20 to 26] | 21.5 [20 to 24] | 24 [21 to 35.5] | 22 [20.5 to 25.5] | 21.5 [20.5 to 24.5] | 22 [20 to 26]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 8 | 8 | 8 | 40
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 8 | 8 | 8 | 40
Serum FSH [Median (Inter-Quartile Range); unit: IU/L] — serum follicle-stimulating hormone
  IU/L | 2.3 [1.5 to 3.5] | 2.7 [1.8 to 3.0] | 2.7 [2.3 to 2.9] | 2.4 [1.7 to 2.8] | 2.3 [1.4 to 3.0] | 2.6 [1.7 to 3.0]
Serum Testosterone [Median (Inter-Quartile Range); unit: ng/mL] | 5.5 [5.2 to 6.2] | 5.4 [4.4 to 6.4] | 5.2 [4.6 to 6.3] | 5.3 [4.7 to 6.3] | 5.2 [4.2 to 5.8] | 5.3 [4.8 to 6.2]
Serum DHT [Median (Inter-Quartile Range); unit: ng/mL] | 0.44 [0.35 to 0.54] | 0.5 [0.43 to 0.89] | 0.5 [0.37 to 0.59] | 0.44 [0.35 to 0.53] | 0.42 [0.3 to 0.5] | 0.46 [0.36 to 0.56]
Serum E2 [Median (Inter-Quartile Range); unit: pg/mL] | 39 [16.5 to 65.8] | 24 [20.9 to 30] | 28.3 [21.3 to 39.6] | 39 [23.4 to 69.4] | 39.4 [21.1 to 51.2] | 28.3 [20.9 to 53.9]
Serum ADD [Median (Inter-Quartile Range); unit: ng/mL] — Serum androstenedione
  ng/mL | 0.7 [0.57 to 1.1] | 0.75 [0.5 to 1.1] | 0.76 [0.52 to 1.12] | 0.69 [0.59 to 0.76] | 0.65 [0.6 to 0.81] | 0.67 [0.57 to 0.95]
Serum DHEA [Median (Inter-Quartile Range); unit: ng/mL] — serum dehydroepiandrosterone
  ng/mL | 3.9 [2.7 to 7.1] | 3.9 [3.2 to 6.6] | 4.2 [3.3 to 6.5] | 4.6 [2.8 to 5.9] | 3.8 [2.8 to 4.4] | 3.9 [2.9 to 6.1]
Serum 17-OHP [Median (Inter-Quartile Range); unit: ng/mL] — serum 17-hydroxyprogesterone
  ng/mL | 6 [4.2 to 7.9] | 6.1 [5.1 to 9.1] | 7.2 [5.9 to 9.5] | 4.8 [4.2 to 6.7] | 6 [4.6 to 9] | 6.1 [4.7 to 8.1]
Serum LH [Median (Inter-Quartile Range); unit: IU/L] — serum luteinizing hormone
  IU/L | 5 [3.1 to 6.6] | 4.7 [4.2 to 5.4] | 4.3 [3.3 to 5.2] | 5.8 [4.7 to 7.4] | 4.9 [4.2 to 6.6] | 4.8 [3.9 to 6.4]

OUTCOME MEASURES:

1. Primary Outcome: Intratesticular Testosterone (IT-T) Level
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Acyline + Testosterone Gel + Placebo: 300mcg Acyline, 1% testosterone gel 5g daily + placebo
- Acyline + Tgel + Ketoconazole 400mg: 300mcg Acyline, 1% testosterone gel 5g daily + 400 mg ketoconazole
- Acyline + Tgel + Ketoconazole 800mg: 300mcg Acyline, 1% testosterone gel 5g daily + 800 mg ketoconazole
Arm/Group | Acyline + Testosterone Gel + Placebo | Acyline + Tgel + Ketoconazole 400mg | Acyline + Tgel + Ketoconazole 800mg | Acyline & TGel & Dutasteride 2.5mg | Acyline & TGel & Anastrazole 1mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng/mL | 14 [8 to 21.2] | 3.7 [2.6 to 7.2] | 1.7 [0.9 to 4] | 18.4 [15.3 to 24.8] | 24.0 [17.7 to 42]
Statistical Analysis 1: Comparison: Acyline + Testosterone Gel + Placebo vs Acyline + Tgel + Ketoconazole 400mg vs Acyline + Tgel + Ketoconazole 800mg vs Acyline & TGel & Dutasteride 2.5mg vs Acyline & TGel & Anastrazole 1mg; Test type: Non-Inferiority or Equivalence — 80% power to detect 20% difference in ITT; p < 0.05, Kruskal-Wallis

2. Primary Outcome: Intratesticular Dihydrotestosterone (DHT) Level
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Acyline + Testosterone Gel (Tgel)+ Placebo: Acyline 300mcg/kg Subcutaneous (SC) (day 1) + testosterone Gel 5g daily x10 days + placebo
- Acyline & TGel & Ketoconazole 400 mg: Acyline 300mcg/kg Subcutaneous (SC) (day 1) + testosterone Gel 5g daily x10 days + ketoconazole 400mg x 7 days
- Acyline & TGel & Ketoconazole 800 mg: Acyline 300mcg/kg Subcutaneous (SC) (day 1) + testosterone Gel 5g daily x10 days + 800mg ketoconazole x 7 days
- Acyline & TGel & Dutasteride: Acyline 300mcg/kg Subcutaneous (SC) (day 1) + testosterone Gel 5g daily x10 days + dutasteride 2.5mg x 7 days
- Acyline & TGel & Anastrazole: Acyline 300mcg/kg Subcutaneous (SC) (day 1) + testosterone Gel 5g daily x10 days + Anastrazole 1mg x 7 days
Arm/Group | Acyline + Testosterone Gel (Tgel)+ Placebo | Acyline & TGel & Ketoconazole 400 mg | Acyline & TGel & Ketoconazole 800 mg | Acyline & TGel & Dutasteride | Acyline & TGel & Anastrazole
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng/mL | 3.17 [2.18 to 3.9] | 2.08 [1.55 to 2.35] | 1.46 [0.75 to 2.25] | 0.12 [0.09 to 0.15] | 3.63 [1.47 to 4.16]
Statistical Analysis 1: Comparison: Acyline + Testosterone Gel (Tgel)+ Placebo vs Acyline & TGel & Ketoconazole 400 mg vs Acyline & TGel & Ketoconazole 800 mg vs Acyline & TGel & Dutasteride vs Acyline & TGel & Anastrazole; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

3. Primary Outcome: Intratesticular Androstenedione (ADD) Level
Time Frame: 10 days
Measure: Median (Inter-Quartile Range); unit: ng/mL
Groups:
- Acyline + Tgel + Ketoconazole 400mg; Acyline + Tgel + Ketoconazole 800mg: Acyline injection 300 mcg/kg SC (day 1) + Testosterone gel 5g + ketoconazole
Arm/Group | Acyline + Testosterone Gel (Tgel)+ Placebo | Acyline + Tgel + Ketoconazole 400mg | Acyline + Tgel + Ketoconazole 800mg | Acyline & TGel & Dutasteride 2.5mg | Acyline & TGel & Anastrazole 1mg
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 8
ng/mL | .87 [.67 to 2.1] | 0.5 [0.3 to 0.7] | 0.12 [0.1 to 0.5] | 1.7 [1.14 to 3.0] | 3.6 [1.6 to 11.9]
Statistical Analysis 1: Comparison: Acyline + Testosterone Gel (Tgel)+ Placebo vs Acyline + Tgel + Ketoconazole 400mg vs Acyline + Tgel + Ketoconazole 800mg vs Acyline & TGel & Dutasteride 2.5mg vs Acyline & TGel & Anastrazole 1mg; Test type: Superiority or Other; p < 0.05, Kruskal-Wallis

ADVERSE EVENTS:
Arm/Group | Acyline & T Gel & Ketoconazole 400 | Acyline & T Gel & Dutasteride | Acyline & T Gel & Placebo Ketoconazole | Acyline & T Gel & Ketoconazole 800 | Group 5: Anastrazole
Serious Adverse Events (participants affected / at risk) | 1/8 | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/8 | 2/8 | 5/8 | 6/8 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyline & T Gel & Ketoconazole 400 (N=8) | Acyline & T Gel & Dutasteride (N=8) | Acyline & T Gel & Placebo Ketoconazole (N=8) | Acyline & T Gel & Ketoconazole 800 (N=8) | Group 5: Anastrazole (N=8)
Testicular hematoma and hematocele (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Development of testicular hematoma and scrotal hematocele after second testicular aspiration on day 10. Underwent operative evacuation of hematocele and cauterization of superficial testicular vessel. Follow-up ultrasound showed complete recovery
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acyline & T Gel & Ketoconazole 400 (N=8) | Acyline & T Gel & Dutasteride (N=8) | Acyline & T Gel & Placebo Ketoconazole (N=8) | Acyline & T Gel & Ketoconazole 800 (N=8) | Group 5: Anastrazole (N=8)
abdomenal ecchymosis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Change in mood/irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased libido (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Finger laceration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
Pain at spermatic cord/at scrotum (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
platar fascitis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergies (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
pruritus/rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No